CLINICAL TRIAL: NCT03814603
Title: A Single-center, Observational, Longitudinal Study on the Effect of Slow Wave Sleep (SWS) Characteristics and Race and Ethnicity on Amyloid Burden (a Marker of Alzheimer's Disease Risk), Among Cognitively Normal Elderly
Brief Title: The Sleep Amyloid, Slow WAve Race and Ethnicity Study
Acronym: Sleep AWARE
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: s18-01302
Record Dates: First submitted 2018-12-27; First posted 2019-01-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood will be drawn for clinical labs and to obtain DNA for ApoE genotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African Americans
  Interventions: Procedure: PET-MR Scan; Drug: PiB
- Non-Hispanic Whites
  Interventions: Procedure: PET-MR Scan; Drug: PiB

INTERVENTIONS:
Procedure: PET-MR Scan — Participants will undergo PET-MR scans at baseline and two-year follow up to examine brain amyloid deposition longitudinally.
Drug: PiB — Subjects will receive a single dose of 555 MBq of PiB and perform a dynamic 30 min PiB PET-MR scan 60 min after injection.

SUMMARY:
African-Americans (AAs) have an increased prevalence of both Alzheimer's disease (AD) and vascular risk factors for AD such as diabetes and hypertension when compared to whites. However, in a recent community based study of non-demented elderly, black race was associated with higher amyloid burden after adjusting for vascular risk factors, suggesting the presence of additional physiological differences on AD-risk by race in the early stages of the disease. The purpose of this study is to test whether poor slow wave sleep (SWS) quantity (SWS duration) and quality (slow wave activity, SWA) is one of these physiological factors. To test these hypotheses, the investigators will perform community outreach in churches and community-based organizations in Brooklyn and other NYC boroughs with which we have created substantial ties in recent years. In consultation with community stakeholders, the investigators will recruit 150 cognitively normal AA elderly (age 60-75) and 60 age, sex, BMI, income and education matched non-Hispanic whites from the same geographical areas. Investigators will first perform a medical and cognitive evaluation (Visit 1). Participants will then undergo 2 nights of home sleep monitoring using an unattended device to exclude OSA, followed by 7 days of actigraphy with a sleep log to record sleep duration. Both devices will be returned by mail. Subjects with reported total sleep time (TST) between 5 and 10 hours and absence of moderate to severe OSA will be invited to perform a 2-night nocturnal polysomnography (NPSG) (Nights 1-2) and a PiB-PET MR scan (Visit 2).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with normal cognition and ages 60 to 75.
* Within normal limits on neurological and psychiatric examinations. All subjects enrolled will have a CDR=0.
* An informed family member or life-partner (preferably bed-partner) will be interviewed over the phone or on the first or second visit to confirm the reliability of the subject interview. A study partner is preferably a spouse, close friend, or relative.
* Self-identified as African-American Black or non-Hispanic white.
* All subjects must sign the Alzheimer's Disease Center consent form

Exclusion Criteria:

* History of brain tumor, MRI evidence of brain damage or brain disease including significant trauma, hydrocephalus, seizures, mental retardation or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders).
* Significant history of alcoholism based off of the CAGE questionnaire (>2) or drug abuse.
* History of psychiatric illness (e.g., schizophrenia, bipolar or PTSD)
* Lifelong depression and anxiety will be allowed as long as there has been no active depressive episode within the last two years.
* Geriatric Depression Scale (short form)>6.
* Insulin dependent diabetes.
* Evidence of clinically relevant cardiac, pulmonary, endocrine or hematological conditions based off of the PI's discretion.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
* Medications affecting cognition or SWS:

  * Narcotic analgesics.
  * Chronic use of medications with anticholinergic activity.
  * Anti-Parkinsonian medications (carbidopa/levodopa, amantadine, bromocriptine, pergolide, selegiline).
  * Others: amphetamines, amphetamine-like compounds, appetite suppressants, phenothiazines, reserpine, buspirone, clonidine, disulfiram, guanethidine, MAO inhibitors, theophylline, tricyclic antidepressants, gabapentin, pregabalin, trazodone, cholinesterase inhibitors, memantine.
* Chronic use of antidepressants are allowed.
* History of a first-degree family member with early onset (age <60 years) dementia.
* Short sleepers (< 5 hours a day) and long sleepers (> 10 hours a day).
* OSA (defined as AHI4%>15 and AHI4%>5 with Epworth≥10)
* Self-identified as US-born Caribbean Black, Caribbean-born Black or African-born Black.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 210 cognitively normal elderly (Clinical Dementia Rating [CDR]=0), self-identified as African-American (AA) or non-Hispanic white (NHW), ages 60 to 75 years, with English as their primary language
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Association between Percentage of African Ancestry (%AF) and Slow Wave Sleep (SWS) duration and activity (SWA). | Determined at baseline.
  Aim 1 will test if individual % African ancestry (%AF), estimated from 0-100 and computed using a maximum likelihood method for inferring individual admixture based upon allele frequencies ascertained from Utah residents with Northern and Western European ancestry and West African samples, is associated with short SWS duration/ and poor slow wave activity (SWA), determined through polysomnography, in older AAs while controlling for other moderating factors.
Examine association between SWS duration and poor SWA with longitudinal change in amyloid burden. | Baseline and 2.5 year follow-up
  Aim 2 will test the effect of race and its interaction with baseline SWS duration and SWA with amyloid plaque burden both at baseline and follow-up by determining mean PiB standard uptake value using PET-MR.
Examine the association between race, SWS duration and poor SWA and cognition using both standardized and sleep-dependent cognitive tests at baseline and follow-up. | Baseline and 2.5 year follow-up
  Aim 3 will test the effect of race and baseline SWS duration and poor SWA on overall cognition using standardized and sleep-dependent tests: the UDS 3.0, WHICAP Clinical Core Neuropsychological test battery, as well as a 3-D Virtual Maze Task, both at baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio, MD, Principal Investigator — NYU Department of Psychiatry
Locations (1):
- NYU Center for Brain Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Subjects will have the option to allow their leftover blood and DNA samples to be banked indefinitely for future research related to studies on early diagnosis of Alzheimer's, disease and/or mechanism of neurodegeneration. After the study is completed, the de-identified, archived data will be transmitted to and stored at the CBH Biorepository, under the supervision of Dr. Osorio, for use by other researchers including those outside of the study. Permission to transmit data to the CBH Biorepository will be included in the ICF. During the conduct of the study, an individual participant can choose to withdraw consent to have biological specimens stored for future research. However, withdrawal of consent with regard to biosample storage will not be possible after the study is completed. When the study is completed, access to study data and/or samples will be provided through the CBH Biorepository.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT03814603/Prot_SAP_000.pdf